CLINICAL TRIAL: NCT01840436
Title: A Randomized Controlled Study Evaluating the Effect of MUCIPLIQ Versus Placebo on the Incidence of Radio-chemotherapy-induced Mucositis in Patients Suffering of Upper Aerodigestive Tract Carcinomas
Brief Title: Efficacy of MUCIPLIQ on the Incidence of Radio-chemotherapy-induced Mucositis in Patients Suffering From Oral Cancer
Acronym: MUCIPLIQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organ, Tissue, Regeneration, Repair and Replacement (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT11M10MURT
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Oral Mucositis; Carcinoma in Situ of Upper Respiratory Tract
Keywords: MUCIPLIQ; Matrix therapy; RGTA; Oral mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): This arm receives a placebo (saline solution) mouthwash treatment twice a day.
  Interventions: Device: Placebo
- MUCIPLIQ 0.05 mg/mL (Experimental): This arm receives MUCIPLIQ mouthwash treatment at a final concentration of 0.05 mg/mL twice a day.
  Interventions: Device: MUCIPLIQ
- MUCIPLIQ 0.015 mg/mL (Experimental): This arm receives MUCIPLIQ mouthwash treatment at a final concentration of 0.015 mg/mL twice a day.
  Interventions: Device: MUCIPLIQ

INTERVENTIONS:
Device: MUCIPLIQ — MUCIPLIQ is applied by mouthwash, for 2 to 3 minutes before being spat out, twice a day.
  Arms: MUCIPLIQ 0.015 mg/mL; MUCIPLIQ 0.05 mg/mL
Device: Placebo — Placebo is applied by mouthwash, for 2 to 3 minutes before being spat out, twice a day.
  Arms: Placebo

SUMMARY:
MUCIPLIQ is a nanopolymer engineered to mimic glycosaminoglycans such as heparan sulfates. Glycosaminoglycans are involved 1) in the stabilization of cells micro-environment, known as extracellular matrix, by binding to structural proteins, and 2) in cells communication process by protecting growth factors. At the site of a lesion, glycosaminoglycans are degraded, thereby the extracellular matrix is disorganized and the tissue is destroyed. By replacing damaged glycosaminoglycans, MUCIPLIQ provides a protection, and restores the matrix scaffold and cells communication, a process known as Matrix Therapy.

The purpose of this new controlled study is to determine whether MUCIPLIQ can decrease the incidence and the severity of radio-chemotherapy-induced mucositis in patients suffering of upper aerodigestive tract cancers, when used as a preventive agent.

The study's main hypothesis is that MUCIPLIQ mouthwash applications before radiotherapy would protect the healthy oral tissue against cytotoxic effect of chemotherapy and radiations.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from an upper aerodigestive tract carcinoma treated by radiotherapy alone or radiotherapy associated with a concomitant platine-salts-based chemotherapy ;
* Patient suffering of an upper aerodigestive tract carcinoma without entrance or located in the oral cavity, in the oropharynx or in the rhinopharynx ;
* Patient age of 18 years old or higher ;
* Writing informed consent to participate to the trial ;
* Patient affiliated to the French social security system.

Exclusion Criteria:

* Treatment by non-standard fragmentation (concentrate irradiation)
* Carcinoma located in the hypopharynx or in the larynx ;
* Known hypersensitivity to heparinoids ;
* Patient who already benefited from a radiotherapy treatment ;
* Patient who already benefited from a chemotherapy treatment. Patients who benefited from neoadjuvant chemotherapy as part of their upper aerodigestive tract carcinoma care, may be included if it was held at least 4 weeks before the inclusion visit ;
* Patient participating to another biomedical research ;
* Pregnant woman, breastfeeding woman, parturient or likely to be ;
* Patient deprived of freedom, under supervision or guardianship ;
* Patient unable to attend to scheduled medical monitoring due to geographical, social or mental reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 2 or higher oral mucositis | Recruitment, 2, 3, 4, 5, 6, 7 and 11 to 13 weeks
  Differences of incidence of patients suffering of oral mucositis of grade 2 or higher

SECONDARY OUTCOMES:
Number and Terms of grade 2 or higher oral mucositis | Recruitment, 2, 3, 4, 5, 6, 7 and 11 to 13 weeks
  Differences of number and terms of oral mucositis of grade 2 or higher between MUCIPLIQ and placebo groups
Administered-antalgics posology and nature | Recruitment, 2, 3, 4, 5, 6, 7 and 11 to 13 weeks
  Differences of administered-antalgics posology and nature between MUCIPLIQ and placebo groups
Pain experienced in time | Recruitment, 2, 3, 4, 5, 6, 7 and 11 to 13 weeks
  Differences of pain experienced by patients between MUCIPLIQ and placebo groups, assessed with Numerical Pain Scale (0 to 10).
Assessment of the Oral Health Impact Profile | Recruitment, 2, 3, 4, 5, 6, 7 and 11 to 13 weeks
  Assessment of the Oral Health Impact Profile assessed by the OHIP-14 questionnaire between MUCIPLIQ and placebo groups
Weight curve | Recruitment, 2, 3, 4, 5, 6, 7 and 11 to 13 weeks
  Assessment of the weight curves for MUCIPLIQ and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Daly-Schveitzer, MD, PhD, Principal Investigator — Institut Gustave Roussy, Villejuif, France; Yungan Tao, MD, Principal Investigator — Institut Gustave Roussy, Villejuif, France; Denis BARRITAULT, PhD, Study Director — Organ, Tissue, Regeneration, Repair and Replacement
Locations (5):
- France (5):
  - Centre de Cancérologie Léon Bérard, Lyon
  - CHRU de Besançon, Site du CH Belfort-Montbéliard, Montbéliard
  - Centre Hospitalier Intercommunal de Créteil, Créteil, Île-de-France Region
  - APHP - Hôpital Tenon, Paris, Île-de-France Region
  - Institut de Cancérologie Gustave Roussy, Villejuif, Île-de-France Region